CLINICAL TRIAL: NCT01938807
Title: Audio Health Engagement Analysis in Diabetes: The AHEAD Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UCSF 12-09213
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; parents; mobile application; diabetes management
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group receives the CareCoach mobile application
  Interventions: Behavioral: CareCoach mobile application to assist in diabetes management
- Control (Active Comparator): The control group receives standard care.
  Interventions: Behavioral: CareCoach mobile application to assist in diabetes management

INTERVENTIONS:
Behavioral: CareCoach mobile application to assist in diabetes management

SUMMARY:
Despite multidisciplinary care and advancements in therapeutics and technology, health outcomes remain suboptimal in pediatric diabetes centers world-wide. A major contributor to poor outcomes is suboptimal diabetes management in pediatric patients and their families. The premise of this research project is that patients and families do not have adequate resources to meet the level of diabetes management that translates to better outcomes. Therefore, we will give them a valuable tool to improve their overall management. The tool is CareCoach.

Research shows that enhancing communication and partnership among patients, parents, and providers is especially critical for optimal outcomes in pediatric diabetes. Communication gaps and conflict can complicate the already complex provider-patient interactions and daily management. We have therefore designed, refined, and made available to consumers a new mobile-based intervention, CareCoach, to improve communication; build trust among providers, patients and parents; and increase overall satisfaction with the quality of diabetes care. This web/mobile application is designed to help patients unobtrusively audio record their clinical encounters, track their medical consults and treatment plans, review information from past visits, create visit discussion guides, and track adherence to medication and dosing schedules. In addition, because mobile-based applications are inexpensive to administer, portable, and available at all times of day, CareCoach holds great promise for communication coaching and contributing to improved diabetes management.

We hypothesize that CareCoach will improve patient-parent-provider communications, build patient-parent-provider trust, and increase overall satisfaction with clinical interactions in a sample of children with type 1 diabetes and their parents. These improvements will lead to significant gains in diabetes management, setting the stage for optimal health outcomes. To test the effectiveness of CareCoach, we will conduct a randomized controlled trial comparing the CareCoach intervention to standard care in a sample of 60 children with type 1 diabetes and their parents.

ELIGIBILITY:
Inclusion Criteria:

* parent of a child with diagnosis of type 1 diabetes for at least one year
* parent of a child with type 1 diabetes between the ages of 7-12
* provide informed consent in English
* have access to the internet from home

Exclusion Criteria:

* no access to the internet
* shorter duration of type 1 diabetes than one year

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09-29 (Actual); Study Completion 2015-09-29 (Actual)

PRIMARY OUTCOMES:
Diabetes Management | 6 months post-baseline

SECONDARY OUTCOMES:
Hemoglobin A1c | 6 months post-baseline

OTHER OUTCOMES:
Satisfaction and usability of the mobile application | 6 months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Diana Naranjo, PhD, Principal Investigator — University of California, San Francisco